CLINICAL TRIAL: NCT04108143
Title: Use of MonitorMe in COPD: a Mixed-methods Feasibility Study
Brief Title: Use of MonitorMe in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: Sanandco Ltd (Unknown); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 181003
Record Dates: First submitted 2019-09-03; First posted 2019-09-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Telehealth; Telemonitoring; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): MonitorMe device
  Interventions: Device: MonitorMe

INTERVENTIONS:
Device: MonitorMe — MonitorMe replaces the users existing telephone and for the majority of time is used as their ordinary telephone. At a known and set time of day for 4 weeks, participants will receive an automated MonitorMe telephone call. The participant answers a health and well-being automated script by pressing key pad numbers. At the same time vital signs data are collected. The responses and vital signs data, together with confidence values are then transmitted via telephone lines to an electronic patient record.

SUMMARY:
MonitorMe is a telephone device intended for the non-critical monitoring of vital signs in a domestic environment with the ability to automatically transmit data to a remote location via basic telephone connectivity.

MonitorMe's low-cost, call automation and simple to use technology (i.e. based on the principles of an ordinary plug-in telephone) make it appropriate for a wide number of care pathways. It eliminates the need for a modem or broadband and avoids the challenges of less reliable smart phone technology. Typical use scenarios include remote monitoring of individual or multiple chronic disease states such as COPD to improve patient outcomes including prevention of emergency admissions.

There is growing interest in the use of home telemonitoring in COPD in order to facilitate the management of the increasing numbers of patients and pressures on the NHS. Despite the positive effects of telemonitoring in conditions such as heart failure, benefits remain unproven in COPD and further work is required before wide-scale use.

Furthermore, until now the evaluation of telecare and telehealth developments has focused mainly on effectiveness and efficiency, whereas their social, and ethical implications in particular, have not been explored in depth. We will also explore ethical issues related to the use of telehealth systems, from both the patients' and the healthcare professionals' perspective.

The current feasibility study is designed to assess the acceptability, usability and validity of MonitorMe within one of its intended purposes i.e. remote monitoring of individual or multiple chronic disease states such as COPD.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Adults diagnosed with any severity of COPD (according to British Thoracic Society criteria, i.e. >10 pack year smoking history and post bronchodilator spirometry FEV1/FVC ratio <0.70 and FEV<80%)
* Listed on referral lists or COPD registers within Lincolnshire Community Health Services NHS Trust or NHS South West Lincolnshire CCG

Health care professionals

* Involved in implementing the device within Lincolnshire Community Health Services NHS Trust or NHS South West Lincolnshire CCG
* Provide informed consent to participate in an interview

Exclusion Criteria:

Patients

* Inability or unwillingness to sign informed consent
* No active telephone line in home
* COPD exacerbation within the previous 6 weeks.
* Mental health, cognitive or neurological conditions that would make study participation inappropriate
* Life expectancy < 6 months
* Implanted pacemaker
* Hearing or visual ailments that would preclude the use of the MonitorMe device
* Inability to use both hands (i.e. hold handset in one hand and use keypad with the other at same time)
* Inability to understand verbal English

Health care professionals

* Not involved in implementing the device within Lincolnshire Community Health Services NHS Trust or NHS South West Lincolnshire CCG
* Unable/unwilling informed consent to participate in an interview

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | Day 0 to 28
  Agreement between measurements made by MonitorMe and healthcare professionals

SECONDARY OUTCOMES:
Temperature | Day 0 to 28
  Agreement between measurements made by MonitorMe and healthcare professionals
Heart rate/pulse rate | Day 0 to 28
  Agreement between measurements made by MonitorMe and healthcare professionals
Adverse event rate | Day 0 to 28
  Number of reported adverse events during study period
Patient compliance | Day 0 to 28
  Number of MonitorMe automated calls completed during observation period
Usability | Day 0 to 28
  Number of unsuccessful data transmissions or missing data (confidence values of MonitorMe)
Acceptance/experience of MonitorMe for patients | Day 28 to 84
  Semi-structured interviews
Acceptance/experience of MonitorMe for health care professionals | Day 28 to 84
  Semi-structured interviews
Self-reported disease specific assessment of quality of life | Day 0 and Day 28
  Chronic Respiratory Questionnaire
Recruitment rates | 1 year
  Time taken to achieve planned sample size
Consent rate | 1 year
  Number of eligible patients willing to consent to take part in the study
Retention rate | Day 0 to 28
  Number of patients who complete the study

CONTACTS AND LOCATIONS:
Overall Officials: Aloysius N Siriwardena, MBBS, PhD, Principal Investigator — University of Lincoln
Locations (2):
- United Kingdom (2):
  - University of Lincoln, Lincoln
  - Lincolnshire Community Health Services NHS Trust, Lincoln

IPD SHARING:
Plan to Share IPD: No